CLINICAL TRIAL: NCT06338449
Title: The Impact of Different Exercise Modes on Bile Acid Levels and Liver Function in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Yang Qiang, Associate professor, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XZMU-2022-ZK068
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD
Keywords: non-alcoholic fatty liver disease; aerobic exercise; resistance exercise; bile acids; liver function
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The specific exercise plan and grouping are as follows:
  Participants were randomly (Using an electronic random number generator) divided into four groups: control group (Control), aerobic training group (AT), resistance training group (RT), and combined aerobic and resistance training group (AT + RT), with each group consisting of 10 individuals, totaling 40 participants. All participants were young adults aged between 18 and 21 years old.
Who Masked: Outcomes Assessor
Masking Description: After the data is obtained, the person analyzing the data will not know the specific grouping and participant information. The groups will be replaced by Group A, B, C, D, and the participants will be indicated by their IDs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic training (AT) (Active Comparator): Aerobic exercise can include activities like swimming, running, or cycling. Scientifically, aerobic exercise is defined as any activity that uses large muscle groups, can be maintained continuously, and is rhythmic in nature. It improves the efficiency of the cardiovascular, respiratory, and circulatory systems by delivering oxygen more efficiently to the body. According to reports, aerobic exercise can help reduce fat and improve liver function.
  Interventions: Behavioral: Aerobic training (AT)
- Resistance training (RT) (Active Comparator): Resistance exercise is a form of physical activity that is designed to improve muscular fitness by exercising a muscle or a muscle group against external resistance. This includes traditional weightlifting, using weight machines, resistance band exercises, bodyweight exercises, and other activities designed to build muscle strength, endurance, and size. The key principle is the muscle's ability to contract against resistance: using weights, resistance bands, or one's own body weight, the muscle is challenged, leading to muscular adaptation and growth, enhancing strength and endurance. According to reports, resistance exercise can also help improve liver function.
  Interventions: Behavioral: Resistance training (RT)
- Combined aerobic and resistance training (AT + RT) (Active Comparator): The combination of aerobic exercise and resistance exercise.
  Interventions: Behavioral: Combined aerobic and resistance training (AT + RT)

INTERVENTIONS:
Behavioral: Aerobic training (AT) — An exercise program was developed by a full-time physical education teacher, with all group exercises conducted at the outdoor track and field facility of Xuzhou Medical University. Participants in the aerobic training group, after completing a warm-up, were required to perform moderate-intensity aerobic running for 60 minutes per session, 4-5 times a week. The exercise intensity was set to reach 50%-70% of the maximum heart rate (Maximum heart rate = 220 - age). The exercise sessions were scheduled in the evening after dinner, from 17:30 to 19:00.All participants were continuously intervened for 8 weeks.
  Arms: Aerobic training (AT)
Behavioral: Resistance training (RT) — Participants in the resistance training group were required to complete moderate-intensity resistance exercises 4-5 times per week. Each session included a warm-up, followed by exercises such as knee lifts with torso twists, knee-to-hand taps under the hips, jumping jacks, burpees, sit-ups, planks, and squats. The routine was structured to perform 5-6 exercises per session, with 6-8 repetitions for each set. There was a 30-second rest interval between sets, and the total exercise time was 60 minutes. The timing for these exercise sessions was the same as for the AT group, conducted in the evening after dinner.All participants were continuously intervened for 8 weeks.
  Arms: Resistance training (RT)
Behavioral: Combined aerobic and resistance training (AT + RT) — Participants in the combined aerobic and resistance training (AT+RT) group started their sessions with a warm-up, followed by 30 minutes of aerobic running. After the aerobic training, they engaged in resistance training. The resistance training regimen was the same as that for the RT group, except that the duration of the resistance training was shorter. The total duration of the exercise session was 60 minutes.All participants were continuously intervened for 8 weeks.
  Arms: Combined aerobic and resistance training (AT + RT)

SUMMARY:
The purpose of this clinical trial is to investigate which exercise regimen is more effective in improving non-alcoholic fatty liver disease (NAFLD) in a young population. The primary questions it aims to answer are:

Does aerobic training, resistance training, or a combination of both help improve liver function and glycemic and lipid parameters in NAFLD patients? Which of these three exercise regimens is more effective in improving the aforementioned parameters? Is the improvement in liver function related to bile acid metabolism?

Participants will:

Engage in physical exercise 4-5 times per week for two consecutive months, following a predefined exercise regimen.

Have blood samples collected to test for glucose, lipids, liver function, and other parameters before starting the exercise program and after two months of completing the regimen.

ELIGIBILITY:
Inclusion Criteria:

* Body fat percentage >20% or BMI >24
* The diagnostic result of abdominal ultrasonography is fatty liver
* No regular exercise under guidance in the past 3 months
* No medication taken in the last month
* No binge eating or heavy drinking in the past two weeks

Exclusion Criteria:

* Long history of alcohol consumption, equivalent to more than 30g/day of ethanol
* Viral hepatitis
* History of autoimmune or genetic diseases
* History of drug-induced liver disease
* History of total parenteral nutrition
* History of cardiovascular, respiratory, or other diseases that necessitate avoidance of intense physical activity.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in body weight compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in Body Mass Index compared to baseline at 8 weeks | Baseline and 8 weeks
  BMI
Changes in total cholesterol compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in triglycerides compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in high-density lipoprotein compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in low-density lipoprotein compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in alanine aminotransferase compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in aspartate aminotransferase compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in alkaline phosphatase compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in gamma-glutamyl transferase compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in direct bilirubin compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in total bile acids compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in adenosine deaminase compared to baseline at 8 weeks | Baseline and 8 weeks

SECONDARY OUTCOMES:
Changes in percentage of body fat compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in waist-to-hip ratio compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in blood glucose compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in the level of insulin compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in albumin compared to baseline at 8 weeks | Baseline and 8 weeks
Changes in C-reactive protein compared to baseline at 8 weeks | Baseline and 8 weeks

OTHER OUTCOMES:
Changes in other subtypes of bile acids compared to baseline at 8 weeks | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Outdoor track and field facility of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The experimental data involves personal privacy and will only be publicly shared when necessary.

REFERENCES:
- [Derived] Shi J, Cui J, Zheng T, Han X, Wang B, Wang W, Zhu C, Fang C, Zhou X, Cong N, Yin X, Yang Q. Comparative effects of aerobic and resistance exercise on bile acid profiles and liver function in patients with non-alcoholic fatty liver disease. BMC Gastroenterol. 2025 Apr 10;25(1):239. doi: 10.1186/s12876-025-03826-x. PMID 40211236